CLINICAL TRIAL: NCT00174304
Title: An International, Multicentre, Open Label Study To Assess The Effectiveness Of Amlodipine/Atorvastatin Combination In Subjects With Hypertension And Dyslipidaemia. (The JEWEL II Study)
Brief Title: Open Label Study To Assess The Effectiveness Of Amlodipine-Atorvastatin Combination In Hypertension And Dyslipidemia.
Acronym: JEWEL II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3841029
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Amlodipine

INTERVENTIONS:
Drug: Amlodipine/atorvastatin single pill

SUMMARY:
To evaluate the effectiveness of amlodipine/atorvastatin therapy by assessing the percentage of subjects who reach target blood pressure (BP) and LDL-C targets as defined by their governing guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Treated or untreated subjects with concurrent hypertension and dyslipidemia with BP and LDL-C not at target according to governing guidelines

Exclusion Criteria:

* High liver enzymes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120
Dates: Start 2004-10; Study Completion 2006-09

PRIMARY OUTCOMES:
To evaluate the effectiveness of amlodipine/atorvastatin therapy by assessing percentage of subjects who reach target BP and LDL-C targets as defined by their governing guidelines.

SECONDARY OUTCOMES:
To asses changes since baseline of lab parameters, BP, safety of titration of amlodipine.atorvastatin to reach targets, to validate Expectations and Satisfaction with Treatment questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- Austria (4):
  - Pfizer Investigational Site, Salzburg
  - Pfizer Investigational Site, Sankt Pölten
  - Pfizer Investigational Site, Vienna
  - Pfizer Investigational Site, Wels
- Belgium (9):
  - Pfizer Investigational Site, Bierbeek
  - Pfizer Investigational Site, Braine-l'Alleud
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, De Pinte
  - Pfizer Investigational Site, GozÃ©e
  - Pfizer Investigational Site, Seraing
  - Pfizer Investigational Site, Wemmel
  - Pfizer Investigational Site, Wilrijk
  - Pfizer Investigational Site, Zedelgem
- Finland (6):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
  - Pfizer Investigational Site, Vantaa
- Greece (8):
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Ioannina
  - Pfizer Investigational Site, Larissa
  - Pfizer Investigational Site, Melíssia
  - Pfizer Investigational Site, Pireaus
  - Pfizer Investigational Site, Rio, Patra
  - Pfizer Investigational Site, Thessaloniki
- Hungary (7):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, KecskemÃ©t
  - Pfizer Investigational Site, Miskolc
  - Pfizer Investigational Site, MosonmagyarÃ³vÃ¡r
  - Pfizer Investigational Site, PÃ©cs
  - Pfizer Investigational Site, SzekszÃ¡rd
- Ireland (2):
  - Pfizer Investigational Site, Gorey, Wexford
  - Pfizer Investigational Site, New Ross, Wexford
- Italy (27):
  - Pfizer Investigational Site, Vimercate, (MI)
  - Pfizer Investigational Site, Somma Lombardo, (VA)
  - Pfizer Investigational Site, San Sisto, PG
  - Pfizer Investigational Site, Mestre, VE
  - Pfizer Investigational Site, Asti
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Bolzano
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Chieti
  - Pfizer Investigational Site, Ferrara
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Grosseto
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Novara
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Potenza
  - Pfizer Investigational Site, Prato
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Salerno
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Venezia
- Portugal (9):
  - Pfizer Investigational Site, Guilhufe - PNF, Penafiel
  - Pfizer Investigational Site, Matosinhos Municipality, Sra. Da Hora
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Faro
  - Pfizer Investigational Site, Leiria
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, S. Martinho Do Bispo
  - Pfizer Investigational Site, Viana do Castelo
- Slovenia (3):
  - Pfizer Investigational Site, Izola
  - Pfizer Investigational Site, Ljubljana
  - Pfizer Investigational Site, Maribor
- Spain (4):
  - Pfizer Investigational Site, Donostia / San Sebastian, Guipuzcoa
  - Pfizer Investigational Site, Reus, Tarragona
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- Switzerland (7):
  - Pfizer Investigational Site, Baden, Canton of Aargau
  - Pfizer Investigational Site, Basel, Canton of Basel-City
  - Pfizer Investigational Site, Bern, Canton of Bern
  - Pfizer Investigational Site, Sankt Gallen, Canton of St. Gallen
  - Pfizer Investigational Site, Lausanne, Canton of Vaud
  - Pfizer Investigational Site, Lugano, Canton Ticino
  - Pfizer Investigational Site, MÃ¼nsterlingen, Thurgau
- Pfizer Investigational Site

REFERENCES:
- [Derived] Richard Hobbs FD, Gensini G, John Mancini GB, Manolis AJ, Bauer B, Genest J, Feldman RD, Harvey P, Jenssen TG, da Silva PM; JEWEL Study Group. International open-label studies to assess the efficacy and safety of single-pill amlodipine/atorvastatin in attaining blood pressure and lipid targets recommended by country-specific guidelines: the JEWEL programme. Eur J Cardiovasc Prev Rehabil. 2009 Aug;16(4):472-80. doi: 10.1097/HJR.0b013e32832b63f5. PMID 19407658
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841029&StudyName=Open+Label+Study+To+Assess+The+Effectiveness+Of+Amlodipine%2DAtorvastatin+Combination+In+Hypertension+And+Dyslipidemia%2E